CLINICAL TRIAL: NCT05569486
Title: Elucidating the Central Mechanism(s) of Action for Green Light Therapy in Managing Chronic Pain
Brief Title: Elucidating the Central Mechanisms of Action for Green Light Therapy in Managing Chronic Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Banner Alzheimer's Institute (Other)
Responsible Party: Principal Investigator, Mohab Ibrahim, PhD MD, Associate Professor, Anesthesiology, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00000333
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Green light-emitting diode (GLED) (Experimental): Subjects randomized to this arm will be exposed to GLED 2 hours a day for 10 weeks
  Interventions: Device: Green Light
- White light-emitting diode (WLED) (Placebo Comparator): Subjects randomized to this arm will be exposed to WLED 2 hours a day for 10 weeks
  Interventions: Device: Green Light

INTERVENTIONS:
Device: Green Light — This is a low-energy device. It produces almost no heat because it uses an LED source for light. The device does not store energy or electrical power that can be discharged later.

SUMMARY:
Investigators have previously shown that specific colors of light can alter nociception. Green light emitting diode exposure (GLED) provides long-lasting antinociception in rodents, through the visual system. No adverse effects were noted, and motor performance was not impaired. Investigator clinical trials have shown GLED is also effective in decreasing pain intensity of fibromyalgia patients and decreasing the number of headache-days per month in migraine patients. However, investigators do not yet understand the mechanisms by which GLED reduces pain.

Understanding the mechanisms of action of GLED will provide additional support for using light therapy as both a treatment and as a possible diagnostic tool. While investigators do not fully understand the mechanisms of action of GLED, investigators do know that it is centrally mediated.

To better elucidate the mechanism of action for GLED, investigators propose a single-blinded randomized placebo-controlled clinical trial to elucidate the central mechanism(s) of action that GLED therapy has in improving fibromyalgia pain, conducted by a team with a successful record of collaboration. Investigator's hypothesis is that GLED decreases neuroinflammation leading to modulation of the signaling in the ascending and descending pain pathways.

DETAILED DESCRIPTION:
After a patient is consented, investigators will collect the baseline Fibromyalgia Impact Questionnaire survey (FIQ), thermal and mechanical pain detection and tolerance threshold, conditioned pain modulation (CPM), collect cerebrospinal fluid (CSF), and obtain positron emission tomography scan (PET scan) for microglia baseline activity. It is expected that the PET scan will take place on different day given the time needed and preparation for the completion of a PET scan. Investigators expect the baseline value collections to take 1-2 days to complete. Once all baseline values are obtained, the light therapy exposure will begin. The start of light exposure will be considered the start of Week 1. Investigators will follow up with the patient over the phone every 2 weeks +/- 1 week to ensure safety and compliance and to answer any questions the patient may have. Recruited patients will also have investigator's contact information to contact investigators with any urgent questions. At the end of Week 10, investigators will obtain the final values for the FIQ survey, thermal and mechanical pain detection and tolerance threshold, CPM, collect CSF, and obtain PET scan.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older who can speak and understand English
* Meets the diagnostic criteria for fibromyalgia accroding to the 2016 revisions to the 2010/2011 fibromyalgia diagnostic criteria.
* Average numeric pain score of 5 out of 10 or greater over the 10 weeks prior to enrolling in the study, and failure of medical therapy to control their pain.

Exclusion Criteria:

* Serious mental illness defined as distortions of perception, delusions, hallucinations, and unusual behaviors resulting in loss of contact with reality. This will be assessed during the screening interview. Patients with psychiatric disorders will have their medical record reviewed prior to enrollment
* History of color blindness or uncorrected cataracts
* Subjects receiving remuneration for their medical condition.
* Genotype of low affinity binders for translocator protein, (TSPO), as patients with low affinity binding TSPO may not have adequate uptake for the radioactive tracer used for the PET scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Decreased activation of glial cells. | [Time Frame: 10 - 22 weeks, depending on study arm]
  By exposure to GLED investigators hypothesize that glial cells will be decreased, investigators will measure this by using positron emission tomography (PET) scan, scans will be conducted at baseline and the end of study

SECONDARY OUTCOMES:
Decreasing Central Nervous System inflammation (CNS), Increasing Endorphins. | [Time Frame: 10 - 22 weeks, depending on study arm]
  By exposure to GLED, investigators hypothesize that inflammation in the CSF will be decreased and increased endorphin levels, this will be demonstrated by measuring cerebrospinal fluid (CSF) cytokines at baseline and at the end of study.
Decreasing the activity of ascending pain pathway, and increasing the activity the descending pain pathway | [Time Frame: 10 - 22 weeks, depending on study arm]
  Decreasing the activity of the ascending pain pathway shown by decreased pain scores from repeated noxious stimulation (temporal summation) as compared to baseline, increasing the activity of the descending pain pathway measured by increasing the pain threshold to noxious stimulation while patients submerge their hand in an ice water bath as compared to baseline.
Improvement in Fibromyalgia Impact Questionnaire score | [Time Frame: 10 - 22 weeks, depending on study arm]
  These will be completed at baseline and at the end of study. A survey to evaluate the effects of Fibromyalgia. The scale ranges from 0-100. 0 means no impact. 100 means there is a severe negative impact secondary to fibromyalgia. The scale is subjective in nature.
Decreased objective and subjective pain scores to mechanical and thermal stimulation | [Time Frame: 10 - 22 weeks, depending on study arm]
  Investigators will compare pain scores at baseline to end of study. The scale ranges from 0-100%. This is a reported value by the patient which is subjective in nature.

CONTACTS AND LOCATIONS:
Overall Officials: Mohab M Ibrahim, PhD., MD, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center Multispecialty Services Clinic, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burckhardt CS, Clark SR, Bennett RM. The fibromyalgia impact questionnaire: development and validation. J Rheumatol. 1991 May;18(5):728-33. PMID 1865419
- [Background] Potvin S, Marchand S. Pain facilitation and pain inhibition during conditioned pain modulation in fibromyalgia and in healthy controls. Pain. 2016 Aug;157(8):1704-1710. doi: 10.1097/j.pain.0000000000000573. PMID 27045524
- [Background] Overstreet DS, Michl AN, Penn TM, Rumble DD, Aroke EN, Sims AM, King AL, Hasan FN, Quinn TL, Long DL, Sorge RE, Goodin BR. Temporal summation of mechanical pain prospectively predicts movement-evoked pain severity in adults with chronic low back pain. BMC Musculoskelet Disord. 2021 May 10;22(1):429. doi: 10.1186/s12891-021-04306-5. PMID 33971876
- [Background] Mackey IG, Dixon EA, Johnson K, Kong JT. Dynamic Quantitative Sensory Testing to Characterize Central Pain Processing. J Vis Exp. 2017 Feb 16;(120):54452. doi: 10.3791/54452. PMID 28287532
- [Background] Yarnitsky D, Bouhassira D, Drewes AM, Fillingim RB, Granot M, Hansson P, Landau R, Marchand S, Matre D, Nilsen KB, Stubhaug A, Treede RD, Wilder-Smith OH. Recommendations on practice of conditioned pain modulation (CPM) testing. Eur J Pain. 2015 Jul;19(6):805-6. doi: 10.1002/ejp.605. Epub 2014 Oct 20. PMID 25330039
- [Background] Yarnitsky D, Granot M, Nahman-Averbuch H, Khamaisi M, Granovsky Y. Conditioned pain modulation predicts duloxetine efficacy in painful diabetic neuropathy. Pain. 2012 Jun;153(6):1193-1198. doi: 10.1016/j.pain.2012.02.021. Epub 2012 Apr 3. PMID 22480803